CLINICAL TRIAL: NCT03802344
Title: A Randomised, Multicentre, Investigator-Blind, Parallel-Group Trial to Evaluate the Efficacy and Safety of MC2-01 Cream Compared to Vehicle and Active Comparator in Subjects With Mild-to-Moderate Psoriasis Vulgaris
Brief Title: This Trial is a Randomised, Multicentre, Investigator-blind, Vehicle and Comparator-controlled, Parallel-group Trial With the Purpose of Evaluation Efficacy, Safety and Convenience of the MC2-01 Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC2-01-C7
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MC2-01 Cream (Experimental): MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0,005%/0,064%) cream. One application daily for 8 weeks
  Interventions: Drug: MC2-01 cream
- Cal/BDP combination (Active Comparator): Calcipotriene/betamethasone (Calcipotriene/betamethasone dipropionate, w/w 0,005%/0,064%) cream. One application daily for 8 weeks
  Interventions: Drug: Cal/BDP combination
- Vehicle (Placebo Comparator): One application daily for 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: MC2-01 cream — MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0,005%/0,064%) cream
  Arms: MC2-01 Cream
Drug: Cal/BDP combination — Calcipotriene/betamethasone dipropionate, w/w 0,005%/0,064%
  Arms: Cal/BDP combination
Drug: Vehicle — Vehicle cream
  Arms: Vehicle

SUMMARY:
This trial is a randomized, investigator-blind, multicentre, vehicle- and comparator-controlled, parallel-group trial with the purpose of evaluating the efficacy, safety and convenience of the MC2-01 cream.

DETAILED DESCRIPTION:
The MC2-01 Cream is designed for optimal patient satisfaction - it quickly absorbs into the skin leaving it nicely moisturized allowing patients to move on in daily routines. In this trial, the MC2-01 cream will be compared to a marketed product CAL/BDP combination and vehicle. The purpose of the trial is to compare the clinical efficacy, safety, and convenience of this cream to the marketed product. The trial will include a 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Generally healthy males or non-pregnant females, of any race or ethnicity, who are at least 18 years of age at the time of screening
* Have a clinical diagnosis of plaque psoriasis (psoriasis vulgaris) of at least 6 months duration that involves the body (trunk and/or limbs) that is amenable to topical treatment with a maximum of 15 g of trial medication per day
* Have a PGA of disease severity of mild or moderate on the body (trunk and/or limbs)
* Have an mPASI score of at least 3
* Have a treatment area involving 2-30% of the body (trunk and/or limbs). For subjects with scalp psoriasis included in the treatment area, the total treatment area on body and scalp must not exceed 30%.

Exclusion Criteria:

* Current diagnosis of unstable forms of psoriasis
* Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris
* Presence of pigmentation, extensive scarring, pigmented lesions or sunburn in the treatment areas
* Planned excessive or prolonged exposure to either natural or artificial sunlight
* History of hypersensitivity to any component of the test product or reference product
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders
* Systemic treatment with biological therapies
* Use of systemic treatments that suppress the immune system and other systemic chemotherapeutic antineoplastic therapy within 4 weeks prior to Visit 1/Baseline and during the trial
* Use of phototherapy within 4 weeks prior to Visit 1/Baseline and during the trial
* Use of topical treatments except for emollients and non-medicated shampoos, with a possible effect on psoriasis within 2 weeks prior to Visit 1/Baseline
* Presence of infections in the treatment area (bacteria, viruses, parasites or fungi) or skin manifestations of atrophic skin, atrophic striae, skin vein fragility, ichthyosis, acne vulgaris, acne rosacea, rosacea, ulcers and wound in the treatment area
* Known Human Immunodeficiency Virus (HIV) infection
* Have any chronic or acute medical condition that may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial
* Initiation of, or expected changes to, concomitant medication that may affect psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Dermatovenerologie a korektivní dermatologie, Prague, Czechia
- University Medical Center Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Pinter A, Galvan J, Freischlager F. Best Responders and Super-Responders to Calcipotriol and Betamethasone Dipropionate PAD-Cream: A Post Hoc Pooled Analysis of Two Phase 3 Trials. Dermatol Ther (Heidelb). 2025 Jun;15(6):1441-1453. doi: 10.1007/s13555-025-01418-x. Epub 2025 Apr 24. PMID 40274711
- [Derived] Stein Gold L, Pinter A, Armstrong A, Augustin M, Arenberger P, Bhatia N, Praestegaard M, Iversen L, Reich A. Calcipotriene and Betamethasone Dipropionate PAD-Cream Demonstrates Greater Treatment Efficacy in Patients with Moderate-to-Severe Psoriasis Compared to Topical Suspension/Gel: A Subgroup Analysis of Two Phase 3 Studies. Dermatol Ther (Heidelb). 2023 Sep;13(9):2031-2044. doi: 10.1007/s13555-023-00979-z. Epub 2023 Jul 25. PMID 37490268
- [Derived] Praestegaard M, Steele F, Crutchley N. Polyaphron Dispersion Technology, A Novel Topical Formulation and Delivery System Combining Drug Penetration, Local Tolerability and Convenience of Application. Dermatol Ther (Heidelb). 2022 Oct;12(10):2217-2231. doi: 10.1007/s13555-022-00794-y. Epub 2022 Sep 1. PMID 36050567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 12-Dec-2018. Last Subject Last Visit: 02-Oct-2019.
Pre-assignment Details: Prior to randomization, the subject entered a washout period (if required) where anti-psoriatic treatment and other relevant medication/treatments were discontinued as defined by the exclusion criteria. The washout/screening period could last for up to 30 days, depending on which disallowed treatments the subject received.
  498 subjects signed the Informed consent form, 490 subjects were randomized and randomly assigned into 3 treatment groups (MC2-01 cream, active comparator, MC2-01 vehicle).
Groups:
- Vehicle: One application daily for 8 weeks
  Vehicle: Vehicle
Period: Overall Study
Arm/Group | MC2-01 Cream | Cal/BDP Combination | Vehicle
Started | 213 | 209 | 68
Completed | 205 | 203 | 55
Not Completed | 8 | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC2-01 Cream | Cal/BDP Combination | Vehicle | Total
Number analyzed (Participants) | 213 | 209 | 68 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.7) | 51.5 (14.8) | 50.8 (13.1) | 50.2 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 96 | 22 | 195
  Male | 136 | 113 | 46 | 295
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 213 | 209 | 68 | 490
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 211 | 205 | 65 | 481
  Race: Black or African American | 0 | 0 | 2 | 2
  Race: Asian | 1 | 2 | 0 | 3
  Race: Gipsy | 1 | 1 | 0 | 2
  Race: North African | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Czechia | 64 | 63 | 20 | 147
  Germany | 94 | 90 | 30 | 214
  Poland | 55 | 56 | 18 | 129
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Patients were classified in accordance with the following classification: I (pale white skin, blue/hazel eyes, blond/red hair; II (fair skin, blue eyes); III (darker white skin); IV (Light brown skin); V (brown skin); VI (dark brown or black skin)
  Participants
    I | 6 | 2 | 0 | 8
    II | 104 | 103 | 29 | 236
    III | 77 | 76 | 25 | 178
    IV | 20 | 19 | 9 | 48
    V | 6 | 7 | 5 | 18
    VI | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in mPASI (Modified Psoriasis Area and Severity Index) Score
Description: The extent and severity of the participant's psoriasis is assessed using a modified PASI scoring system (minus scalp, face, and flexures) at each 3 areas (arms, trunk and legs) using a scale from 0 - 6, where 0 = no psoriasis involvement and 6 = 90-100% involvement.
  The severity is assessed at the 3 areas for each of the sign redness, thickness and scaliness using a scale from 0 - 4, where 0 represents none and 4 represents very severe.
  The mPASI score is calculated from the individual scores by use of the following equation:
  Arms 0.2 (Redness + Thickness + Scaliness) E = X Trunk 0.3 (Redness + Thickness + Scaliness) E = Y Legs 0.4 (Redness + Thickness + Scaliness) E = Z The sum of X + Y + Z = m-PASI score resulting in a minimum score of 0 and a maximum score (worst possible) of 64.8.
  The percent change in mPASI score is defined as the Baseline minus the Week 8 divided by Baseline score multiplied by 100 (if a reduction is seen the value will be presented as a negative number)
Time Frame: 8 Weeks
Population: The analysis was based on the FAS population.
Measure: Mean (Standard Error); unit: Percentage change from Baseline
Arm/Group | MC2-01 Cream | Cal/BDP Combination | Vehicle
Number analyzed (Participants) | 213 | 209 | 68
Percentage change from Baseline | -67.5 (20.8) | -63.5 (22.2) | -11.7 (21.9)

2. Secondary Outcome: The Psoriasis Treatment Convenience Scale (PTCS)
Description: PTCS measures the impact and convenience of the treatment. The scale consists of 6 disease-specific questions, which individually will be rated on a 1-10 points scale, where a score of 1 represents the lowest satisfactory response with the treatment and 10 represents the highest satisfactory response. The questions are: Q1. How easy was the treatment to apply to the skin?; Q2. How greasy was the treatment when applying it to the skin?; Q3. How moisturized did your skin feel after apolying the treatment?; Q4. How greasy did your skin feel after applying the treatment?; Q5. How much did treating you skin disrupt your daily routine?; Q6. Overall, how satisfied were you with the medical treatment? The total PTCS score is calculated as the sum of the first 5 questions, ranging from 5 [low satisfaction] to 50 [high satisfaction].
Time Frame: 8 Weeks
Population: The analysis was based on the FAS population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MC2-01 Cream | Cal/BDP Combination | Vehicle
Number analyzed (Participants) | 213 | 209 | 68
score on a scale | 38.6 (6.2) | 36.1 (7.0) | 36.2 (7.6)

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time of the signature of the informed consent form by the subject and until the end of the trial, i.e. until the Follow-up visit at Week 10. AEs that were considered related to the trial product would be followed until they were resolved, or until the medical condition of the subject was stable.
Arm/Group | MC2-01 Cream | Cal/BDP Combination | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/209 | 0/68
Serious Adverse Events (participants affected / at risk) | 1/213 | 3/209 | 1/68
Other Adverse Events (participants affected / at risk) | 10/213 | 11/209 | 1/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-01 Cream (N=213) | Cal/BDP Combination (N=209) | Vehicle (N=68)
Testicular seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholesystitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-01 Cream (N=213) | Cal/BDP Combination (N=209) | Vehicle (N=68)
Nasopharyngitis (Infections and infestations) | 10 (10) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03802344/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03802344/SAP_001.pdf